CLINICAL TRIAL: NCT06051253
Title: Efficacy of Infliximab Treatment Based on TDM (Therapeutic Drug Monitoring) in Adult Patients With Active Perianal Fistulizing Crohn's Disease
Brief Title: TDM-based Infliximab Treatment for Active Perianal Fistulizing Crohn's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Byong Duk Ye, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220573
Record Dates: First submitted 2023-09-10; First posted 2023-09-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Crohn Disease; Infliximab; Perianal Fistula Due to Crohn's Disease; Therapeutic Drug Monitoring; Magnetic Resonance Novel Index for Fistula Imaging in Crohn's Disease Score
MeSH Terms: conditions — Crohn Disease | interventions — CT-P13

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDM-based group (Experimental): At week 0,2, and 6, infliximab (CT-P13, RemsimaTM) is intravenously administered at a dose of 5 mg/kg. From week 14 to 46 (at week 14, 22, 30, 38, and 46), infliximab dose can be increased to 10 mg/kg, targeting trough level (TL) of infliximab 10 mcg/mL or over (If TL is 10 mcg/mL or over under treatment with 5 mg/kg infliximab, 5 mg/kg of infliximab is continued. If TL is lower than 10 mcg/mL, infliximab dose is increased to 10 mg/kg). Once infliximab dose was increased to 10 mg/kg, the next doses are fixed to 10 mg/kg.
  Interventions: Drug: TDM-based infliximab intravenous therapy
- Standard group (Active Comparator): Infliximab (CT-P13, RemsimaTM) is intravenously administered at a dose of 5 mg/kg at week 0, 2, 6, 14, 22, 30, 38, and 46. Therapeutic dose monitoring (TDM, checking trough levels of infliximab) is performed at week 14, 22, 30, 38, and 46, but TDM results are not reflected in determining doses of infliximab.
  Interventions: Drug: Standard infliximab intravenous therapy

INTERVENTIONS:
Drug: TDM-based infliximab intravenous therapy — Infliximab (CT-P13, RemsimaTM) is intravenously given as an induction therapy at a dose of 5 mg/kg at week 0, 2, and 6. From week 14 to 46 (at week 14, 22, 30, 38, and 46), infliximab dose can be increased to 10 mg/kg, targeting trough level (TL) of infliximab 10 mcg/mL or over (If TL is 10 mcg/mL or over under treatment with 5 mg/kg infliximab, 5 mg/kg of infliximab is continued. If TL is lower than 10 mcg/mL, infliximab dose is increased to 10 mg/kg). Once infliximab dose was increased to 10 mg/kg, the next doses are fixed to 10 mg/kg.
  Other Names: TDM-based infliximab (CT-P13, RemsimaTM) intravenous therapy
  Arms: TDM-based group
Drug: Standard infliximab intravenous therapy — Infliximab (CT-P13, RemsimaTM) is intravenously administered at a dose of 5 mg/kg at week 0, 2, 6, 14, 22, 30, 38, and 46. Therapeutic dose monitoring (TDM, checking trough levels of infliximab) is performed at week 14, 22, 30, 38, and 46, but TDM results are not reflected in determining doses of infliximab.
  Other Names: Standard infliximab (CT-P13, RemsimaTM) intravenous therapy
  Arms: Standard group

SUMMARY:
This study will compare the efficacy and safety of TDM (therapeutic drug monitoring)-based infliximab (CT-P13, RemsimaTM) intravenous therapy compared with the standard infliximab (RemsimaTM) intravenous therapy for patients with active perianal fistulzing Crohn's disease.

DETAILED DESCRIPTION:
The TDM-based group: At week 0,2, and 6, infliximab (RemsimaTM) is intravenously administered at a dose of 5 mg/kg. From week 14 to 46 (at week 14, 22, 30, 38, and 46), infliximab dose can be increased to 10 mg/kg, targeting trough level (TL) of infliximab 10 mcg/mL or over (If TL is 10 mcg/mL or over under treatment with 5 mg/kg infliximab, 5 mg/kg of infliximab is continued. If TL is lower than 10 mcg/mL, infliximab dose is increased to 10 mg/kg). Once infliximab dose was increased to 10 mg/kg, the next doses are fixed to 10 mg/kg.

The standard group: Infliximab (RemsimaTM) is intravenously administered at a dose of 5 mg/kg at week 0, 2, 6, 14, 22, 30, 38, and 46. Therapeutic dose monitoring (TDM, checking trough levels of infliximab) is performed at week 14, 22, 30, 38, and 46, but TDM results are not reflected in determining doses of infliximab.

The co-primary endpoints of the study will be 1) Clinical remission (both week 50 and week 54), 2) Changes of MAGNIFI-CD (Magnetic Resonance Novel Index for Fistula Imaging in Crohn's Disease) score compared with the baseline score (week 54)

ELIGIBILITY:
* Inclusion Criteria:

  1. Age: 19-80 years
  2. Subjects diagnosed with perianal fistulizing Crohn's disease based on clinical, endoscopic, histological, and radiologic findings, etc.
  3. Subjects naive to both biological drugs (anti-TNFs, anti-integrin, anti-IL12/23, etc.) and investigational new drugs
  4. Subjects with at least one draining perianal fistula
  5. Subjects not responding to two or more conventional treatments (antibiotics, drainage, immunosuppressants, etc.)
  6. Women with a childbearing potential: Those who agree to follow contraception during study drug administration and for at least 6 months from the last dosing of the study medication
* Exclusion Criteria:

  1. In cases where written informed consents cannot be provided by the study subjects or the subjects' legally acceptable representative
  2. Subject with a probability of receiving bowel surgery within 12 weeks after baseline, decided by investigators
  3. Subjects with temporary or permanent stoma
  4. Subjects with short bowel syndrome
  5. Subjects not eligible due to significant bowel strictures or intra-abdominal abscesses
  6. Subjects who received bowel surgery within 6 months of baseline or subjects who were admitted due to complications associated with bowel strictures or intra-abdominal abscesses within 3 months of baseline
  7. Subjects with enterovaginal fistula, enterocutaneous fistula, or enteroenteric fistula
  8. Subjects previously exposed to biologics (anti-TNFs, anti-integrin, anti-IL12/23, etc.) or investigational new drugs
  9. Subjects with a history of hypersensitivity to monoclonal antibody
  10. Subjects requiring corticosteroid therapy. However, if oral corticosteroid dose lower or equivalent to prednisolone 20 mg/day before baseline is given and tapering of oral corticoseroid from baseline is planned, that subjects can be included in the study. Oral corticoseroid is tapered at a schedule of prednisolone 5 mg/7 days (example: if the subject was on oral prednisolone 20 mg/day before baseline, oral prednisolone is tapered as follows: 15 mg/day x 7 days -> 10 mg/day x 7 days -> 5 mg/day x 7 days -> stopping of prednisolone)
  11. Subjects with active tuberculosis. However, if the subject has a history of tuberculosis, which was cured with standard anti-tuberculosis therapy according to the standard anti-tuberculosis treatment guidelines, that subject can be included
  12. Subjects with latent tuberculosis: Subjects determined to be positive for latent tuberculosis by the pulmonology specialist after history taking, physical examination, chest X-ray, and interferon gamma release assay during the screening period. However, even if positive for latent tuberculosis, if 4 week-treatment for latent tuberculosis is completed and if further treatment for latent tuberculosis is planned to be completed, that subject can be included
  13. Subjects positive for HBsAg. In cases of HBsAg (-), but with IgG Anti-HBc (+), real time quantitative PCR for HBV DNA is required. If HBV DNA is 10 IU/mL or over, that subject should be excluded
  14. Subjects positive for anti-HCV antibody
  15. Subjects with a history of infection with HIV or subject positive for HIV Ag
  16. Subjects positive for Clostridioides difficile toxin assay or Clostridioides difficile culture assay
  17. Subjects with a heart disease of NYHA Class III/IV
  18. Subjects with current or previous demyelinating disease
  19. Subject with a history of malignancy (excluding skin basal cell carcinoma, skin squamous cell carcinoma, and uterine cervix cancer) within 5 years or with a history of dysplasia of colon or small bowel within 5 years.
  20. Subjects with symptoms or signs of active infection or with a history of treatment for infection within 8 weeks
  21. Subjects with a history of organ transplantation
  22. Pregnant or lactating women
  23. Non-Korean ethnicity according to a family tree
  24. Subjects decided to be not eligible for the study by investigators

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants in clinical remission | Both week 50 and 54
  Clinical remission is defined as no draining perianal fistula on gentle finger compression by a surgeon, without a seton. To be classified as clinical remission, participants should show no draining perianal fistula on gentle finger compression by a surgeon, without a seton at both week 50 and week 54.
Change of the MAGNIFI-CD (Magnetic Resonance Novel Index for Fistula Imaging in Crohn's Disease) score | Week 54
  MAGNIFI-CD = 3 x Number of fistula tract (3 levels) + 2 x Hyperintensity of primary tract on post-contrast T1-weighted images (2 levels) + 2 x Dominant feature (3 levels) + 2 x Fistula length (3 levels) + 2 x Extension (3 levels) + 1 x Inflammatory mass (6 levels).
  Range of values: 0 ~ 25 High values mean more active perianal fistula

SECONDARY OUTCOMES:
Proportion of participants in clinical response | Week 54
  Clinical response is defined as 50% or more decrease of the number of draining fistula or of draining amount on gentle finger compression by a surgeon, without a seton.
The proportion of patients with MAGNIFI-CD (Magnetic Resonance Novel Index for Fistula Imaging in Crohn's Disease) score of 0 | Week 54
  MAGNIFI-CD = 3 x Number of fistula tract (3 levels) + 2 x Hyperintensity of primary tract on post-contrast T1-weighted images (2 levels) + 2 x Dominant feature (3 levels) + 2 x Fistula length (3 levels) + 2 x Extension (3 levels) + 1 x Inflammatory mass (6 levels).
  Range of values: 0 ~ 25 High values mean more active perianal fistula
Biochemical remission | Week 54
  The proportion of patients with biochemical remission (CRP [C-reactive protein] < 0.6 mg/dL)
The median level of infliximab | Week 22, 30, 38, 46 and 54
  Infliximab level is measured by the the Quantum Blue® Infliximab assay measure and is expressed as mcg/mL. In each group, infliximab trough levels of week 22, 30, 38, 46 and 54 are summarized and median value with interquartile ranges are calculated. Between two groups, those median values are compared.
Change of IBDQ (Inflammatory Bowel Disease Questionnaire) score | Week 54
  The IBDQ (Inflammatory Bowel Disease Questionnaire) gives a possible score range of 32 to 224, where a higher score indicates better health-related quality of life. IBDQ is measured at week 14 and week 54.
The proportion of patients with safety issues (adverse events) | Week 54
  Comparing the proportions of patients having any adverse events, serious adverse events, serious infections, and all types of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Byong Duk Ye, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JJ, Yang SK, Ye BD, Kim JW, Park DI, Yoon H, Im JP, Lee KM, Yoon SN, Lee H; IBD Study Group of the Korean Association for the Study of the Intestinal Diseases. [Second Korean Guidelines for the Management of Crohn's Disease]. Korean J Gastroenterol. 2017 Jan 25;69(1):29-54. doi: 10.4166/kjg.2017.69.1.29. Korean. PMID 28135790
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Cheon JH, Kim YS, Ye BD, Lee KM, Kim YH, Kim JS, Han DS, Kim WH. Crohn's Disease Clinical Network and Cohort (CONNECT) Study: The First Step Toward Nationwide Multicenter Research of Crohn's Disease in Korea. Intest Res. 2014 Jul;12(3):173-5. doi: 10.5217/ir.2014.12.3.173. No abstract available. PMID 25349589
- [Background] Klag T, Goetz M, Stange EF, Wehkamp J. Medical Therapy of Perianal Crohn's Disease. Viszeralmedizin. 2015 Aug;31(4):265-72. doi: 10.1159/000434664. Epub 2015 Jul 29. PMID 26557835
- [Background] Park EJ, Song KH, Baik SH, Park JJ, Kang J, Lee KY, Goo JI, Kim NK. The efficacy of infliximab combined with surgical treatment of fistulizing perianal Crohn's disease: Comparative analysis according to fistula subtypes. Asian J Surg. 2018 Sep;41(5):438-447. doi: 10.1016/j.asjsur.2017.06.005. Epub 2017 Aug 26. PMID 28851611
- [Background] Yassin NA, Askari A, Warusavitarne J, Faiz OD, Athanasiou T, Phillips RK, Hart AL. Systematic review: the combined surgical and medical treatment of fistulising perianal Crohn's disease. Aliment Pharmacol Ther. 2014 Oct;40(7):741-9. doi: 10.1111/apt.12906. Epub 2014 Aug 13. PMID 25115149
- [Background] Ye BD, Pesegova M, Alexeeva O, Osipenko M, Lahat A, Dorofeyev A, Fishman S, Levchenko O, Cheon JH, Scribano ML, Mateescu RB, Lee KM, Eun CS, Lee SJ, Lee SY, Kim H, Schreiber S, Fowler H, Cheung R, Kim YH. Efficacy and safety of biosimilar CT-P13 compared with originator infliximab in patients with active Crohn's disease: an international, randomised, double-blind, phase 3 non-inferiority study. Lancet. 2019 Apr 27;393(10182):1699-1707. doi: 10.1016/S0140-6736(18)32196-2. Epub 2019 Mar 28. PMID 30929895
- [Background] Present DH, Rutgeerts P, Targan S, Hanauer SB, Mayer L, van Hogezand RA, Podolsky DK, Sands BE, Braakman T, DeWoody KL, Schaible TF, van Deventer SJ. Infliximab for the treatment of fistulas in patients with Crohn's disease. N Engl J Med. 1999 May 6;340(18):1398-405. doi: 10.1056/NEJM199905063401804. PMID 10228190
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485
- [Background] Ordas I, Feagan BG, Sandborn WJ. Therapeutic drug monitoring of tumor necrosis factor antagonists in inflammatory bowel disease. Clin Gastroenterol Hepatol. 2012 Oct;10(10):1079-87; quiz e85-6. doi: 10.1016/j.cgh.2012.06.032. Epub 2012 Jul 17. PMID 22813440
- [Background] Vande Casteele N, Ferrante M, Van Assche G, Ballet V, Compernolle G, Van Steen K, Simoens S, Rutgeerts P, Gils A, Vermeire S. Trough concentrations of infliximab guide dosing for patients with inflammatory bowel disease. Gastroenterology. 2015 Jun;148(7):1320-9.e3. doi: 10.1053/j.gastro.2015.02.031. Epub 2015 Feb 24. PMID 25724455
- [Background] Papamichael K, Rakowsky S, Rivera C, Cheifetz AS, Osterman MT. Association Between Serum Infliximab Trough Concentrations During Maintenance Therapy and Biochemical, Endoscopic, and Histologic Remission in Crohn's Disease. Inflamm Bowel Dis. 2018 Sep 15;24(10):2266-2271. doi: 10.1093/ibd/izy132. PMID 29718327
- [Background] Yarur AJ, Kanagala V, Stein DJ, Czul F, Quintero MA, Agrawal D, Patel A, Best K, Fox C, Idstein K, Abreu MT. Higher infliximab trough levels are associated with perianal fistula healing in patients with Crohn's disease. Aliment Pharmacol Ther. 2017 Apr;45(7):933-940. doi: 10.1111/apt.13970. Epub 2017 Feb 17. PMID 28211593
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Gionchetti P, Dignass A, Danese S, Magro Dias FJ, Rogler G, Lakatos PL, Adamina M, Ardizzone S, Buskens CJ, Sebastian S, Laureti S, Sampietro GM, Vucelic B, van der Woude CJ, Barreiro-de Acosta M, Maaser C, Portela F, Vavricka SR, Gomollon F; ECCO. 3rd European Evidence-based Consensus on the Diagnosis and Management of Crohn's Disease 2016: Part 2: Surgical Management and Special Situations. J Crohns Colitis. 2017 Feb;11(2):135-149. doi: 10.1093/ecco-jcc/jjw169. Epub 2016 Sep 22. PMID 27660342
- [Background] Regueiro M, Mardini H. Treatment of perianal fistulizing Crohn's disease with infliximab alone or as an adjunct to exam under anesthesia with seton placement. Inflamm Bowel Dis. 2003 Mar;9(2):98-103. doi: 10.1097/00054725-200303000-00003. PMID 12769443
- [Background] Yan X, Zhu M, Feng Q, Yan Y, Peng J, Xu X, Xu A, Ran Z. Evaluating the effectiveness of infliximab on perianal fistulizing Crohn's disease by magnetic resonance imaging. Gastroenterol Rep (Oxf). 2019 Feb;7(1):50-56. doi: 10.1093/gastro/goy036. Epub 2018 Oct 24. PMID 30792866
- [Background] Hindryckx P, Jairath V, Zou G, Feagan BG, Sandborn WJ, Stoker J, Khanna R, Stitt L, van Viegen T, Shackelton LM, Taylor SA, Santillan C, Mearadji B, D'Haens G, Richard MP, Panes J, Rimola J. Development and Validation of a Magnetic Resonance Index for Assessing Fistulas in Patients With Crohn's Disease. Gastroenterology. 2019 Nov;157(5):1233-1244.e5. doi: 10.1053/j.gastro.2019.07.027. Epub 2019 Jul 20. PMID 31336124
- [Background] Davidov Y, Ungar B, Bar-Yoseph H, Carter D, Haj-Natour O, Yavzori M, Chowers Y, Eliakim R, Ben-Horin S, Kopylov U. Association of Induction Infliximab Levels With Clinical Response in Perianal Crohn's Disease. J Crohns Colitis. 2017 May 1;11(5):549-555. doi: 10.1093/ecco-jcc/jjw182. PMID 28453755